CLINICAL TRIAL: NCT05958836
Title: Quality of Life and Clinical Outcomes in Patients Treated With Leadless Micra Transcatheter Pacemakers as Compared With Traditional Transvenous Pacemakers
Brief Title: Quality of Life in Patients Treated With Leadless Pacemakers
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MicraQL
Record Dates: First submitted 2023-07-12; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Leadless Micra Transcatheter Pacemaker; Quality of Life

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Micra TPS group
  Interventions: Device: pacemaker
- Traditional PM group

INTERVENTIONS:
Device: pacemaker — Micra TPS or traditional PM group
  Groups: Micra TPS group

SUMMARY:
The study aims to carry out a domestic multi-center, prospective, non-randomized, non-blinded post-approval study to assess health-related QoL between Micra TPS and conventional PM implantation. Meanwhile, pocket and leads related complications would also be evaluated between these two strategies.

ELIGIBILITY:
Inclusion Criteria:

* With an age arranged from 18 to 80 years old;
* Conforming to indication of a pacemaker implantation;
* Life expectancy>1 year;
* Normal cardiac function with preserved LVEF;
* Adequate self-care ability or self-help skills before pacemaker implantation;
* Mentally healthy so as to participate in the quality-of-life assessments;
* Willing to participate in study through consent and willing to undergo study specific required procedures with expectancy of geographically stable for follow up duration.

Exclusion Criteria:

* Subject with indication for ICD/ CRT-P/CRT-D;
* Subject with persistent symptomatic sinus bradycardia;
* Subject has an existing or prior pacemaker, ICD or CRT device implant;
* Subject has unstable angina pectoris or has an acute myocardial infarction (AMI) in the 30 days prior to eligibility assessment;
* Subjects with a mechanical tricuspid valve, implanted vena cava filter, or left ventricular assist device (LVAD);
* Subjects with a life expectancy of less than 12-months;
* Subjects with medical condition which precludes patient from participation in the opinion of the investigator, such as arthritis, lung disease or previous stroke, renal dysfunction, recent major surgery within six months, clinically overt congestive heart failure;
* Pregnant women or breastfeeding women, or women of child bearing potential and who are not on a reliable form of birth regulation method or abstinence;
* Psychological disorders unable to participate in the quality-of-life assessments.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients are eligible if they meet the indication of a single or dual chamber permanent pacemaker. All subjects should fit the following inclusion criteria and disagree with the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 246 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life measured by EQ-5D-5L | 6 Months post implant
  The EQ-5D-5L results shall be collected during study follow up visits
Health-related quality of life measured by NHP (Nottingham Health Profile) | 6 Months post implant
  The NHP results shall be collected during study follow up visits

IPD SHARING:
Plan to Share IPD: No